CLINICAL TRIAL: NCT00872430
Title: Laxative Effectiveness of a Phytotherapeutic Tea: A Randomized Placebo-Controlled Clinical Trial
Brief Title: Laxative Effectiveness of a Phytotherapeutic Tea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Laboratório Klein Ltda. (Unknown)
Responsible Party: Paulo Dornelles Picon, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 02121
Record Dates: First submitted 2008-11-06; First posted 2009-03-31 (Estimated); Results first posted 2009-03-31 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Constipation
Keywords: constipation; RCT; phytotherapy
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo/Laxative tea crossover (Active Comparator): This arm received placebo in the first period and laxative tea in the second period (after washout period of 9 days).
  Interventions: Other: Placebo; Other: Klein Laxative Tea
- Laxative tea/Placebo crossover (Active Comparator): This arm received laxative tea in the first intervention period and placebo in the second intervention period (after washout period of 9 days).
  Interventions: Other: Placebo; Other: Klein Laxative Tea

INTERVENTIONS:
Other: Placebo — In order to produce similar taste and color, 7 drops of caramel color and 10 drops of orange essence were mixed into 1.6 liters of boiling water. The patients received 150 ml of placebo 3 times a day for 5 days.
Other: Klein Laxative Tea — The laxative tea was prepared using 1 gram of grinded plant into 150 ml of water, left under infusion by 5 minutes. Patients received 150 ml of tea 3 times a day for 5 days.
  Other Names: Phytotherapeutic tea; laxative tea

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of a phytotherapeutic laxative tea, composed by Pimpinella anisum, Foeniculum vulgare, Sambucus nigra and Cassia angustifolia, in a randomized crossover placebo-controlled clinical trial in patients with chronic constipation.

DETAILED DESCRIPTION:
The Klein Laxative Tea is a pharmaceutical phytotherapeutic product that's been used for several years in Brazil for the treatment of constipation. This product contains fruit of Pimpinella anisum (green anises), fruit of Foeniculum vulgare (fennel), flowers of Sambucus nigra (elder tree) and flowers of Cassia angustifolia (senna). In spite of the beneficial effects of its components, separately demonstrated in vitro, it never had its effectiveness appraised in a randomized clinical trial.The purpose of this study was to evaluate the efficacy and safety of this product in a randomized crossover placebo-controlled clinical trial. Twenty patients presenting with the criteria of the American Association of Gastroenterology for chronic constipation were included, and concluded a two-phase crossover study. The primary endpoint was the evaluation of the intestinal transit time measured through radiological technique. The secondary endpoints were the number of evacuations, subjective impression of the quality in the intestinal habit, quality of life appraised through WHOQOL-brief and adverse effects.

ELIGIBILITY:
Inclusion criteria:

* patients with 18 to 55 years old with chronic constipation according to the criteria of the American Association of Gastroenterology (AAG);
* patients should present good understanding and collaboration capacity, an not be in use of other medications with effects on the intestinal habit;
* patients with no abnormalities in the exams;
* willing to sign a written informed consent;
* women in fertile age should make use of appropriate anti-conception.

Exclusion Criteria:

* pregnant or breast feeding women;
* patients with history of abuse of alcohol or use of drugs;
* significant or not-controlled disease, except constipation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2002-07; Primary Completion 2002-12 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo D picon, Coordinator, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Picon PD, Picon RV, Costa AF, Sander GB, Amaral KM, Aboy AL, Henriques AT. Randomized clinical trial of a phytotherapic compound containing Pimpinella anisum, Foeniculum vulgare, Sambucus nigra, and Cassia augustifolia for chronic constipation. BMC Complement Altern Med. 2010 Apr 30;10:17. doi: 10.1186/1472-6882-10-17. PMID 20433751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited by the Clinical Research Unit from output clinic at Hospital de Clínicas de Porto Alegre through written announcements attached to panels inside the institution.
Pre-assignment Details: Twenty patients fulfilled elegibility criteria. No patients were excluded after signing informed consent form and randomization.
Groups:
- Placebo First Crossover: Placebo in the first period and laxative tea in the second period (after washout period)
- Laxative Tea First Crossover: Laxative tea in the first period and placebo in the second period (after washout period).
Period: First Intervention
Arm/Group | Placebo First Crossover | Laxative Tea First Crossover
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Placebo First Crossover | Laxative Tea First Crossover
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First Crossover | Laxative Tea First Crossover
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First Crossover | Laxative Tea First Crossover | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Brazil | 10 | 10 | 20

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients With no Evacuation After Each Intervention Period
Description: The number of patients who had not evacuated on day 5 of each intervention period was obtained using questions 1 and 9 of the Scale for Assessment of Constipation Symptoms based on: 1) How many times have you had a bowel movement in the last 24 hours?; 9) Classification of bowel habit on a scale of 1 (terrible) to 5 (excellent).
Time Frame: day 5 and day 19
Measure: Number; unit: participants
Groups:
- Placebo: Placebo administered three times a day in either first intervention period or second intervention period.
- Laxative Tea: Laxative tea administered three times a day in either first intervention period or second intervention period.
Arm/Group | Placebo | Laxative Tea
Number analyzed (Participants) | 20 | 20
participants | 9 | 0
Statistical Analysis 1: Comparison: Placebo vs Laxative Tea; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Primary Outcome: Intestinal Transit Time
Description: Radiologic technique consisting of the ingestion of radiopaque markers, followed by a simple x-ray of the abdomen on day 3 of each intervention period. Standard formula, regarding markers ingested, time of ingestion and markers still present on the colon (counted by radiologist unaware of the treatment allocation), provided transit time.
Time Frame: day 3 and day 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Laxative Tea
Number analyzed (Participants) | 20 | 20
hours | 42.3 (18.86) | 15.66 (9.71)
Statistical Analysis 1: Comparison: Placebo vs Laxative Tea; All data were collected and entered before the opening of the codes of blinding of researchers. We used t test for paired samples and test for repeated measures linear regression for variables with more than two measures.With an improvement of 40% in the tea group and of 20% in the placebo group, with a power (1-ß) of 80% and a alpha error 0.05, it was necessary to include 32 points of comparison, which would be achieved with at least 16 patients, since it's a crossover study; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No